CLINICAL TRIAL: NCT06884202
Title: Clinical Evaluation of Overall Lens Fit of Delefilcon A Contact Lenses of Different Diameters and Base Curves
Brief Title: Evaluation of Delefilcon A Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLU484-P007
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Refractive Errors; Myopia
Keywords: Contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID023681, then LID006961 (Other): Delefilcon A contact lenses with different base curves and diameters worn in Period 1, followed by delefilcon A contact lenses with standard base curves and diameters worn in Period 2. During each period, the contact lenses will be worn bilaterally (in both eyes) for 6 (+2) hours. A one-to-two day washout will separate the wear periods.
  Interventions: Device: Delefilcon A contact lenses with different base curves and diameters; Device: Delefilcon A contact lenses with standard base curves and diameters
- LID006961, then LID023681 (Other): Delefilcon A contact lenses with standard base curves and diameters worn in Period 1, followed by delefilcon A contact lenses with different base curves and diameters worn in Period 2. During each period, the contact lenses will be worn bilaterally (in both eyes) for 6 (+2) hours. A one-to-two day washout will separate the wear periods.
  Interventions: Device: Delefilcon A contact lenses with different base curves and diameters; Device: Delefilcon A contact lenses with standard base curves and diameters

INTERVENTIONS:
Device: Delefilcon A contact lenses with different base curves and diameters — Silicone hydrogel contact lenses for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.
  Other Names: LID023681
Device: Delefilcon A contact lenses with standard base curves and diameters — Silicone hydrogel contact lenses for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.
  Other Names: DAILIES TOTAL1®; LID006961

SUMMARY:
The purpose of the study is to evaluate the lens fit characteristics of delefilcon A contact lenses with different base curves and diameters.

DETAILED DESCRIPTION:
Subjects will be expected to attend 4 office visits for an individual duration of participation of approximately 3 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Successful wearer of spherical soft contact lenses in both eyes for a minimum of 5 days per week and a minimum of 6 hours per day during the past 3 months;
* Able to wear contact lenses within a range of sphere powers from -2.00 and -4.00 diopters (D);
* Best Corrected Visual Acuity (BCVA) (with manifest refraction) better than or equal to 0.10 logarithm Minimum Angle of Resolution (logMAR ) in each eye.

Key Exclusion Criteria:

* Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator;
* History of refractive surgery or plan to have refractive surgery during the study, or irregular cornea in either eye;
* Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher; presence of corneal infiltrates.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Proportion of lenses graded as Acceptably Tight, Optimal Fit, or Acceptably Loose at Dispense in lens movement (overall lens fit) at primary gaze | Day 1 Dispense (Hour 0) of each study lens type worn during the corresponding crossover period
  Lens movement (overall lens fit) will be evaluated by the investigator using a slit lamp with the eye in primary position. Lens movement (overall lens fit) will be graded on a 5-point scale as follows: -2 = unacceptably tight (reduced movement, unacceptable); -1 = Acceptably tight (reduced movement, acceptable); 0 = Optimal fit / movement; +1 = Acceptably loose (excessive movement, acceptable); +2 = Unacceptably loose (excessive movement, unacceptable).
Proportion of lenses graded as Acceptably Tight, Optimal Fit, or Acceptably Loose at Dispense in lens movement (overall lens fit) at peripheral gazes | Day 1 Dispense (Hour 0) of each study lens type worn during the corresponding crossover period
  Lens movement (overall lens fit) will be evaluated by the investigator using a slit lamp with the eye in upward gaze, downward gaze, looking to the left, and looking to the right. Lens movement (overall lens fit) for each gaze will be graded on a 5-point scale as follows: -2 = unacceptably tight (reduced movement, unacceptable); -1 = Acceptably tight (reduced movement, acceptable); 0 = Optimal fit / movement; +1 = Acceptably loose (excessive movement, acceptable); +2 = Unacceptably loose (excessive movement, unacceptable).
Proportion of lenses graded as Optimal Lens Centration or Acceptable Decentration at Dispense in lens position (centration) | Day 1 Dispense (Hour 0) of each study lens type worn during the corresponding crossover period
  Lens position (centration) will be evaluated by the investigator using a slit lamp with the eye in primary position. Lens position (centration) will be graded on a 3-point scale as follows: 0 = Optimal centration; 1 = Acceptable centration; 2 = Unacceptable decentration.
Proportion of lenses graded as Acceptably Tight, Optimal Fit, or Acceptably Loose at 6 Hour Follow-up in lens movement (overall fit) at primary gaze | Day 1, Hour 6 (+2) of each study lens type worn during the corresponding crossover period
  Lens movement (overall lens fit) will be evaluated by the investigator using a slit lamp with the eye in primary position. Lens movement (overall lens fit) will be graded on a 5-point scale as follows: -2 = unacceptably tight (reduced movement, unacceptable); -1 = Acceptably tight (reduced movement, acceptable); 0 = Optimal fit / movement; +1 = Acceptably loose (excessive movement, acceptable); +2 = Unacceptably loose (excessive movement, unacceptable).
Proportion of lenses graded as Acceptably Tight, Optimal Fit, or Acceptably Loose at 6 Hour Follow-up in lens movement (overall fit) at peripheral gazes | Day 1, Hour 6 (+2) of each study lens type worn during the corresponding crossover period
  Lens movement (overall lens fit) will be evaluated by the investigator using a slit lamp with the eye in upward gaze, downward gaze, looking to the left, and looking to the right. Lens movement (overall lens fit) for each gaze will be graded on a 5-point scale as follows: -2 = unacceptably tight (reduced movement, unacceptable); -1 = Acceptably tight (reduced movement, acceptable); 0 = Optimal fit / movement; +1 = Acceptably loose (excessive movement, acceptable); +2 = Unacceptably loose (excessive movement, unacceptable).
Proportion of lenses graded as Optimal Lens Centration or Acceptable Decentration at 6 Hour Follow-up in lens position (centration) | Day 1, Hour 6 (+2) of each study lens type worn during the corresponding crossover period
  Lens position (centration) will be evaluated by the investigator using a slit lamp with the eye in primary position. Lens position (centration) will be graded on a 3-point scale as follows: 0 = Optimal centration; 1 = Acceptable centration; 2 = Unacceptable decentration.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (16):
- United States (16):
  - Kurata Eyecare Center, Los Angeles, California
  - Elsa Pao, OD, Oakland, California
  - Pacific Rims Optometry, San Francisco, California
  - Pearson Research Center, PA, Longwood, Florida
  - Kindred Optics at Maitland Vision, Maitland, Florida
  - Eyeconic Family Eyecare, Dallas, Georgia
  - Dr. Schwartz Optometrist and Associates, Sterling Heights, Michigan
  - Coldwater Vision Research, Coldwater, Mississippi
  - SUNY College of Optometry Clinical Vision Research Center, New York, New York
  - NC Eye Associates, OD, PLLC, Apex, North Carolina
  - See Eye Care Optometry, Charlotte, North Carolina
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Eyecare Professionals, Inc, Powell, Ohio
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - West Bay Eye Associates, Warwick, Rhode Island
  - Southern College of Optometry, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No